CLINICAL TRIAL: NCT04656730
Title: Effect of STW5 (Iberogast ®) and STW5-II (Iberogast N®) on Transit and Tolerance of Intestinal Gas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Collaborators: Bayer Hispania, S.L (Unknown)
Responsible Party: Principal Investigator, Dr. Jordi Serra Pueyo, MD. PH D., Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBO
Record Dates: First submitted 2020-11-13; First posted 2020-12-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Irritable Bowel Syndrome; Functional Dyspepsia
Keywords: Digestive System Diseases; 2. Gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Digestive System Diseases | interventions — iberogast; Exercise

STUDY DESIGN:
Intervention Model Description: To determine the independent effects of STW5 and STW5-II on transit and evacuation of intestinal gas in subjects with functional dyspepsia and irritable bowel syndrome according to Rome IV criteria, measured as ml of gas recovered by a rectal cannula
Who Masked: Participant, Investigator
Masking Description: Experimental group: Study 1: STW5 20 drops TID; Study 2: STW5-II 20 drops TID Control group: Placebo 20 drops TID
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study 1: Experimental: Study 2: Experimental (Experimental): Iberogast® (STW5) or Iberogast® N (STW5-II) 20 drops TID per 14 days
  Interventions: Drug: Iberogast® and Iberogast® N
- Study 1: Comparator Study 2: Comparator (Placebo Comparator): Placebo 20 drops TID per 14 days
  Interventions: Drug: Iberogast® and Iberogast® N

INTERVENTIONS:
Drug: Iberogast® and Iberogast® N — Oral intake of the investigation drug 20 drops three times per day (TID) for 14 days,
  Other Names: active

SUMMARY:
Study to asess the effects of Iberogast® (STW5) and Iberogast® N (STW5-II) in intestinal gas transit and abdominal symptoms of patients suffering from irritable bowel syndrome or functional dyspepsia.

DETAILED DESCRIPTION:
Every day great amounts of gas enter into the intestine from several sources, including air swallowed during meals and gas produced by colonic fermentation by intestinal bacteria.

Recent studies have shown that gastric nutrients delay emptying of gastric gas in healthy subjects, and this effect is exacerbated in patients with functional dyspepsia, leading to a lower tolerance to gastric gas and greater gas-related epigastric symptoms. Likewise, patients with lower functional gut disorders, like irritable bowel syndrome or functional bloating, have an altered transit and evacuation of intestinal gas that is associated to abdominal symptoms. In addition, bloating and abdominal distension are gas-related abdominal symptoms that are common to both upper and lower functional gut disorders, and referred by a majority of patients, as their most bothersome symptoms.

STW5 (Iberogast®) is a medicinal product composed by 9 herbal preparations that has been shown to promote changes in gastric tone, gastrointestinal motility, intestinal inflammation and visceral sensitivity.

Iberogast® is approved in Spain for treatment of gastrointestinal disorders like dyspepsia and gastritis, as well as for symptomatic relief of associated symptoms as epigastric pain, bloating, flatulence, gastrointestinal colics, nausea and epigastric burning sensation (extract from Summary of product characteristics, SmPC) ).

STW5-II (Iberogast N®) is an herbal medicinal preparation consisting of six herbal extracts (Iberis amara whole plant, caraway fruits, liquorice roots, peppermint leaves, lemon balm leaves, and chamomile flowers). It contains an extract combination of Iberis amara as an alcoholic fresh plant extract as well as plant extracts of caraway fruits, liquorice roots, peppermint leaves, lemon balm leaves, and chamomile flowers as alcoholic drug extracts. The preparation contains 31% ethanol.

Iberogast N® was approved in Germany only on 07 Oct 2010 and is indicated for the treatment of functional gastrointestinal diseases like functional dyspepsia (FD) and irritable bowel syndrome (IBS) . It was marketed with only very few packs to keep the license. It is approved for adolescents and adults from the age of 12 years, as for patients below the age of 12 no data are available.

Iberogast N was tested in five controlled clinical trials with a dosage scheme of 3 x 20 drops/day over 4 to 12 weeks.

Efficacy was proven in the indications FD (four studies) and IBS (one study). Approximately 441 participants have been treated with Iberogast N in clinical studies. The analysis of AEs did not lead to any safety signal or concern and supports the favorable benefit risk profile of BAY98-7410 (STW 5-II).

Three subjects from the overall safety population that participated in 6 interventional studies, experienced at least one SAE, including 1 subject of 139 (0.71%) treated with BAY98-7410 (STW 5-II) (female, 43 years old, hospitalized due circulatory problems, treatment was discontinued) and 2 subjects (1.5%) of 133 treated with placebo (1 male, 65 years old, hospitalized due psychiatric disorders triggered by stressful life events, treatment was discontinued; 1 female, 47 years old, diagnosed during hospitalization with anemia, treatment was discontinued). All SAEs were only reported for the interventional study STW5 II/212-D-03-III-V and were assessed as not related to study treatment (Information from Investigator Brochure).

In addition, laboratory investigations of the subjects during the clinical trials gave no evidence for clinically relevant changes caused by treatment with Iberogast N.

Functional gut disorders comprise a large number of chronic medical conditions that may affect all the segments of the gastrointestinal tract, from the esophagus to the anus, characterized by a combination of disturbances including dysbiosis, altered permeability, altered immunological responses and microinflammation, motor and sensory dysfunction, and altered processing of the gut stimuli by the central nervous system. The most prevalent functional gastrointestinal disorders are functional dyspepsia and irritable bowel syndrome. Functional dyspepsia is characterized by symptoms (pain, burning, fullness and early satiety) referred to the epigastrium, whereas irritable bowel syndrome is characterized by abdominal pain and altered bowel habits. In both disorders gas-related abdominal symptoms, like abdominal bloating and distension, are among the most frequently referred symptoms. Treatment of these gas-related abdominal symptoms is often disappointing, and patients are often advised to follow very restrictive diets, like the low-FODMAP diet, to control these symptoms. However, these restrictive diets are not harmless, because they can lead to malnutrition, and to severe alterations of gut microbiota.

Now-to-date, despite the prevalence of gas-related abdominal symptoms in patients with functional gut disorders, and the multitarget effects of the herbal preparation Iberogast, with several mechanisms of action like changes in motility and sensitivity that could act on bloating and gas retention, there are no studies exploring the effects of Iberogast on intestinal gas transit and tolerance in subjects with functional gut disorders. Hence, the aim of the present trial is to determine the effects of Iberogast, and the simplified formula Iberogast N, on intestinal transit and tolerance in subjects with functional dyspepsia and irritable bowel syndrome according to Rome IV criteria, using a methodology for the study of gas transit that has been largely used and validated by the investigation team.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read and signed the institutional review board-approved informed consent form before screening.
2. ≥18 years old.
3. Confirmed irritable bowel syndrome (ibs) or functional dyspepsia (fd) diagnosis per rome iv criteria.
4. Has active symptoms of bloating.
5. Subject must be willing to comply with the protocol.
6. Female subjects who are capable of conceiving must use an acceptable form of contraception in order to participate in the study*. *women of childbearing potential must have a negative pregnancy test prior to randomization into the study and commitment to use at least one of these birth control methods: male or female condom with or without spermicide, cap, hormonal contraception, diaphragm or sponge with or without spermicide, intrauterine device, bilateral tubal occlusion, vasectomized partner, sexual abstinence during the study. based on ich, m3 (r2) 2009 a woman is considered of childbearing potential: fertile, following menarche and until becoming post-menopausal unless permanently sterile. permanent sterilization methods include tubal ligation, hysterectomy, bilateral oophorectomy.

Exclusion Criteria:

1. Presence of any organic gastrointestinal diseases.
2. Subjects with known hypersensitivity to Iberogast or one of the active substances or excipients.
3. One or more medical condition(s), including renal, hepatic, hematologic, endocrinological, neurologic, or immune disease that in the opinion of the Investigator would make the subject an inappropriate candidate for this study.
4. Subjects with impaired liver function tests
5. Malignant disease not in remission.
6. Presence of any active infectious disease.
7. Subjects not willing to stop medications that may interfere with gastrointestinal motility during 48 h previous to the gas infusion tests. These include: bulking agents, laxatives, linaclotide, prokinetics, antidiarrheal or opioids.
8. Known alcohol or drug abuse.
9. Female participants of childbearing potential with a positive pregnancy test, breast feeding, or female participants of childbearing potential without adequate contraception.
10. Subject judged by the investigator or study staff to be unable or unlikely to comply with daily protocol requirements, or study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Transit and evacuation of intestinal gas | Baseline to Day 14
  Colonic gas filling and evacuation (patients with irritable bowel síndrome) and Gastric gas transit (patients with functional dispepsia).
  Primary outcome measures will be evaluated by an infusion machine (to perform gas infusion) and a barostat (to perform gas collection measurement).

SECONDARY OUTCOMES:
Perception of abdominal symptoms | Baseline to Day 14
  To determine the independent effects of STW5 and STW5-II, compared to respective placebos, on subjective perception of abdominal symptoms (measured by a graded symptom scale) in response to colonic gas infusion in subjects with irritable bowel syndrome and functional dyspepsia.
Objective abdominal distension | Baseline to Day 14
  To determine the independent effects of STW5 and STW5-II, compared to respective placebos, on objective abdominal distension (measured in mm by a tape-measure) in response to colonic gas infusion in subjects with irritable bowel syndrome and functional dyspepsia.
Adverse events | Baseline to Day 14
  To determine the adverse events that occur during the study.

CONTACTS AND LOCATIONS:
Overall Officials: JORDI SERRA, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona